CLINICAL TRIAL: NCT00905073
Title: Low Dose Cyclosporin and Methotrexate Therapy in New Onset Diabetes Mellitus
Brief Title: Low Dose Cyclosporin and Methotrexate Therapy in Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Douglas Sobel, Georgetown University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10988
Record Dates: First submitted 2009-05-19; First posted 2009-05-20 (Estimated); Last update posted 2011-04-13 (Estimated); Status verified 2009-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; cyclosporin; methotrexate; renal function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Cyclosporine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cyclosporin+Methotrexate (Experimental): cyclosporin treatment at 7.5 mg/kg/day for 6 weeks and then 4 mg/kg/day for on year and methotrexate 5 mg/kg/day for one year.
  Interventions: Drug: cyclosporin and methotrexate

INTERVENTIONS:
Drug: cyclosporin and methotrexate — cyclosporin 7.5 mg/kg/day for 6 weeks and then 4 mg/kg/day for one year and methotrexate 5 mg/kg/day for one year. After 6 weeks, cyclosporin doses will adjusted to maintain blood cyclo levels to 100-200 ng/ml.

SUMMARY:
The purpose of this study is to determine whether treatment with low dose cyclosporin and methotrexate can inhibit the development of new onset diabetes mellitus

DETAILED DESCRIPTION:
Objective: Although high doses of cyclosporin (cyclo) inhibits the development of type 1 diabetes mellitus, its usefulness is limited by its toxicity. Since methotrexate (mtx) and cyclo synergistically inhibit other disease processes, we hypothesized that low dose cyclo and mtx therapy could safely induce remission.

Research Design and Methods: In an open pilot study, insulin dose and glycemic control will be compared in children with new onset Type 1 diabetes administered cyclo at 7.5 mg/kg/day for 6 weeks and then 4 mg/kg/day and mtx 5 mg/kg/day for one year with control children. After 6 weeks, doses were adjusted to maintain blood cyclo levels to 100-200 ng/ml.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type1 diabetes mellitus and be obtaining insulin therapy for less than 4 weeks

Exclusion Criteria:

* Ketoacidosis
* Body weight over 110% of ideal weight
* Condition where immunosuppression is contraindicated
* Abnormal liver or renal function tests

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 1990-02; Primary Completion 1994-06 (Actual); Study Completion 1994-06 (Actual)

PRIMARY OUTCOMES:
insulin dose | one year

SECONDARY OUTCOMES:
renal function | one year

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Sobel, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States